CLINICAL TRIAL: NCT03331913
Title: The Efficacy and Safety of Botulinum Toxin for the Treatment of Trigeminal Neuralgia: Comparison of Two Different Treatment Methods
Brief Title: Botulinum Toxin for Trigeminal Neuralgia
Acronym: EASTERN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Chuanjie Wu, MD, PhD, The First Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FAHZU-2017-025
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Trigeminal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Botulinum Toxins, Type A; Injections, Intradermal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intradermal / submucosal injection group (Active Comparator): intradermal / submucosal injection at pain area
  Interventions: Drug: Botulinum Toxin type A (intradermal / submucosal injection at pain area)
- intra-masseter injection group (Experimental): intra-masseter injection on the ipsilateral of pain involved
  Interventions: Drug: Botulinum Toxin type A (intra-masseter injection on the ipsilateral of pain involved)

INTERVENTIONS:
Drug: Botulinum Toxin type A (intradermal / submucosal injection at pain area) — Comparison of two different treatment methods of Botulinum Toxin type A for the treatment of trigeminal neuralgia
  Arms: intradermal / submucosal injection group
Drug: Botulinum Toxin type A (intra-masseter injection on the ipsilateral of pain involved) — Comparison of two different treatment methods of Botulinum Toxin type A for the treatment of trigeminal neuralgia
  Arms: intra-masseter injection group

SUMMARY:
Trigeminal neuralgia (TN) is one of the most painful and common types of neuropathic pain encountered by clinicians. It is typically treated pharmacologically with anticonvulsants,but these can be ineffective, or can lose their effectiveness over time.Botulinum toxin type A (BoNT-A) is an exotoxin released by the Gram-positive, anaerobic bacillus Clostridium botulinum that causes flaccid paralysis by blocking neurotransmitter release by axonal terminals. As a contaminant, it is the cause of potentially lethal botulism poisoning; however, as a drug, it has been widely used in the treatment of dystonia, as well as for non-surgical cosmetic treatment. More recently, studies investigating the ability of BoNT-A to treat pain have been increasing. In 2012, the investigators reported the results of a randomized, double-blind, and placebo-controlled trial in which subcutaneous injection of BoNT-A at the site of pain provided long-term effective relief in TN. The investigators noted that adverse effects were mild, as well. Other studies on TN have estimated the effectiveness of BoNT-A treatment in TN to be 47-73%. However, BoNT-A treatment is still ineffective in more than 30% of patients.In this study, the investigators investigate whether different treatment methods have different efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Clinical diagnosis of classical trigeminal neuralgia according to the ICHD III (beta)
* The pain involved the gingiva
* Signed informed consent prior to entering study

Exclusion Criteria:

* comorbid diseases that may be exacerbated by botulinum toxin type A (e.g., myasthenia gravis, motor neuron disease, or Lambert-Eaton syndrome).
* receiving drugs with neuromuscular junction toxicity 1 week before botulinum toxin type A treatment (e.g. quinine, aminoglycosides or penicillamine)
* had an infection of the skin or mucosa at any of the injection sites.
* psychiatric illness.
* malignancy.
* pregnancy or lactation.
* currently participating or previously participated in any investigational drug or device study within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-11-07 (Actual); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Pain relief | 4 weeks
  Pain relief was defined as ≥50% reduction in Visual Analogue Scale score which is an 11 point scale from 0 - 10 with 0 being no headache

SECONDARY OUTCOMES:
Visual Analogue Scale score | 1 week
  Visual Analogue Scale score is an 11 point scale from 0 - 10 with 0 being no headache
Visual Analogue Scale score | 2 weeks
  Visual Analogue Scale score is an 11 point scale from 0 - 10 with 0 being no headache
Visual Analogue Scale score | 3 weeks
  Visual Analogue Scale score is an 11 point scale from 0 - 10 with 0 being no headache
Visual Analogue Scale score | 4 weeks
  Visual Analogue Scale score is an 11 point scale from 0 - 10 with 0 being no headache
Visual Analogue Scale score | 5 weeks
  Visual Analogue Scale score is an 11 point scale from 0 - 10 with 0 being no headache
Visual Analogue Scale score | 6 weeks
  Visual Analogue Scale score is an 11 point scale from 0 - 10 with 0 being no headache
Visual Analogue Scale score | 7 weeks
  Visual Analogue Scale score is an 11 point scale from 0 - 10 with 0 being no headache
Visual Analogue Scale score | 8 weeks
  Visual Analogue Scale score is an 11 point scale from 0 - 10 with 0 being no headache
Visual Analogue Scale score | 9 weeks
  Visual Analogue Scale score is an 11 point scale from 0 - 10 with 0 being no headache
Visual Analogue Scale score | 10 weeks
  Visual Analogue Scale score is an 11 point scale from 0 - 10 with 0 being no headache
Visual Analogue Scale score | 11 weeks
  Visual Analogue Scale score is an 11 point scale from 0 - 10 with 0 being no headache
Visual Analogue Scale score | 12 weeks
  Visual Analogue Scale score is an 11 point scale from 0 - 10 with 0 being no headache
The overall response to treatment on the Patient Global Impression of Change | 8 weeks

OTHER OUTCOMES:
Safety which is assessed by adverse reactions | 12 weeks
  Adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: Chuanjie Wu, MD, Study Chair — Xuanwu Hospital Captial Medical University
Locations (5):
- China (5):
  - Xuanwu Hospital Captial Medical University, Beijing, Beijing Municipality
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Xiangtan Central Hospital, Xiangtan, Hunan
  - Luzhou People's Hospital, Luzhou, Sichuan